CLINICAL TRIAL: NCT01422733
Title: Effect of Longer-term Adrenal Suppression Using Low Dose Hydrocortisone on Androgen Overproduction in Overweight Early Pubertal Girls With Androgen Excess (CBS0004)
Brief Title: Effect of Longer-term Adrenal Suppression Using Low Dose Hydrocortisone on Androgen Overproduction
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study team decided not to pursue this study.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christine Burt Solorzano, Assistant Professor of Pediatrics, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CBS004; CBS004 (Other: University of Virginia)
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Hyperandrogenemia; Obesity; Polycystic Ovary Syndrome
MeSH Terms: conditions — Obesity; Polycystic Ovary Syndrome | interventions — Hydrocortisone; Dexamethasone; Cosyntropin; Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hydrocortisone, dexamethasone, Cosyntropin (ACTH), rhCG (Experimental): 12 weeks hydrocortisone, dexamethasone, and Cosyntropin (ACTH) to perform standardized adrenal stimulation testing; dexamethasone, and rhCG to perform standardized ovarian stimulation testing
  Interventions: Drug: Hydrocortisone; Drug: dexamethasone; Drug: Cosyntropin; Drug: rhCG

INTERVENTIONS:
Drug: Hydrocortisone — 10mg/m2/per day PO at bedtime (X12 weeks)
Drug: dexamethasone — 1 mg PO twice
Drug: Cosyntropin — 250 micrograms IV twice
  Other Names: Tetracosactide
Drug: rhCG — 25 mcg IV twice
  Other Names: (Ovidrel)

SUMMARY:
This study will test whether longer-term suppression of adrenal function can ameliorate androgen (male hormone) overproduction in overweight early pubertal girls with androgen excess. The investigators hypothesize that suppression of nighttime adrenocorticotropin hormone (ACTH) production by 12 weeks of evening oral hydrocortisone administration will improve androgen levels in girls with adrenal androgen overproduction. Specifically, this intervention will improve androgen levels after adrenal stimulation testing with ACTH or ovarian stimulation testing with recombinant human chorionic gonadotropin (rhCG).

ELIGIBILITY:
Inclusion Criteria:

* Overweight(>85th BMI%) females
* Early puberty defined by Tanner 1-2 breast development (expected age range 7-16)
* Hyperandrogenemic (free testosterone greater than 2.5 standard deviations above the mean for normal control subjects of the same Tanner Stage)
* Screening labs within age-appropriate normal range, with the exception of a mildly low hematocrit (see below) and the hormonal abnormalities inherent in obesity which could include mildly elevated luteinizing hormone (LH), lipids, testosterone, prolactin, DHEAS, E2, glucose, and insulin; and decreased follicle-stimulating hormone (FSH) and/or sex hormone-binding globulin (SHBG)

Exclusion Criteria:

* Age < 7 or > 16 y
* Inability to comprehend what will be done during the study or why it will be done
* BMI-for-age < 5th percentile
* Positive pregnancy test or lactation.
* Screening labs outside of age-appropriate normal range (Abnormal laboratory studies will be confirmed by repeat testing to exclude laboratory error)
* Morning cortisol < 5 µg/dL or history of Cushing syndrome or adrenal insufficiency
* History of congenital adrenal hyperplasia or 17-hydroxyprogesterone > 295 ng/dL, which suggests the possibility of congenital adrenal hyperplasia (if postmenarcheal, the 17-hydroxyprogesterone will be collected during the follicular phase, or ≥ 40 days since last menses if oligomenorrheic). NOTE: If a 17-hydroxyprogesterone >295 mg/dL is confirmed on repeat testing, an ACTH-stimulated 17-hydroxyprogesterone <1000 ng/dL will be required for study participation.
* Total testosterone > 150 ng/dL, which suggests the possibility of a virilizing neoplasm
* DHEAS greater than the upper limit of age-appropriate normal range (mild elevations may be seen in polycystic ovary syndrome (PCOS) and adolescent hyperandrogenemia (HA), and elevations < 1.5 times the age-appropriate upper limit of normal will be accepted in these groups)
* Virilization
* Previous diagnosis of diabetes, fasting glucose ≥126 mg/dL, or a hemoglobin A1c ≥6.5%
* Abnormal thyroid stimulating hormone (TSH) for age. Subjects with stable and adequately treated hypothyroidism, reflected by normal TSH values, will not be excluded.
* Abnormal prolactin. Mild elevations may be seen in overweight girls, and elevations <1.5 times the upper limit of normal will be accepted in this group.
* Persistent hematocrit <36% and hemoglobin <12 g/dL. Subjects with a mildly low hematocrit (33-36%) will be asked to take iron in the form of ferrous gluconate for up to 60 days. Subjects weighing ≤ 36 kg will take one 300-325 mg tablet oral ferrous gluconate daily (containing 36 mg elemental iron);subjects weighing >36 kg will take two 300-325 mg tablets oral ferrous gluconate daily (containing 36 mg elemental iron each). They will return to the Clinical Research Unit (CRU) after 30-60 days of iron therapy to have their hemoglobin or hematocrit rechecked and will proceed with the remainder of the study if it is ≥12 g/dL or ≥36%, respectively.
* Persistent liver test abnormalities, with the exception that mild bilirubin elevations will be accepted in the setting of known Gilbert's syndrome. Mild elevations may be seen in overweight girls, so elevations <1.5 times the upper limit of normal will be accepted in this group.
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.)
* Abnormal sodium, potassium, or bicarbonate concentrations, or elevated creatinine concentration (confirmed on repeat)
* No medications known to affect the reproductive system or glucose metabolism can be taken in the 3 months prior to the study. Such medications include oral contraceptive pills, progestins, metformin, glucocorticoids, and psychotropics.

Ages: 7 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Changes in free testosterone or 17-hydroxyprogesterone levels after ACTH and rhCG administration respectively, before and after hydrocortisone administration for 12 weeks | 12 weeks after hydrocortisone administration

SECONDARY OUTCOMES:
Changes in adrenal and ovarian steroid precursors after ACTH and rhCG; body composition via air displacement plethysmography, BMI, and glucose tolerance testing results; baseline and after 12 weeks of hydrocortisone administration | 12 weeks after hydrocortisone administration
Morning cortisol | 72 hours following discontinuation of hydrocortisone

CONTACTS AND LOCATIONS:
Overall Officials: Christine Burt Solorzano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Research in Reproduction, Charlottesville, Virginia, United States